CLINICAL TRIAL: NCT03600220
Title: Effectiveness of Combining Antihypertensive Drugs and Acupuncture on Isolated Systolic Hypertension of Elderly Patients at Home
Brief Title: Exploring the Effect of Combined Chinese and Western Treatment on Home Medical Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Taipei City Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TCHIRB-10703120-E
Record Dates: First submitted 2018-06-25; First posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-06

CONDITIONS: Hypertension
Keywords: acupuncture, hypertension, elderly, home health care
MeSH Terms: conditions — Hypertension | interventions — Acupuncture Therapy; Pharmaceutical Preparations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- drug use (No Intervention): routine drug use, each patient was using 1-3 antihypertensive drug of a heterogeneous pharmacological group ranging from ACE inhibitors, diuretics, and beta blockers
- drug combine acupuncture (Experimental): routine drug use combine acupuncture twice a week for 3 months
  Interventions: Other: acupuncture

INTERVENTIONS:
Other: acupuncture — antihypertension drug, acupuncture twice a week for 3 months
  Other Names: drug
  Arms: drug combine acupuncture

SUMMARY:
combine antihypertensive drugs and acupuncture to isolated systolic hypertension elderly patients at home

DETAILED DESCRIPTION:
The investigators would like to compare the effectiveness of acupuncture and drug therapy on blood pressure.

The investigators chose acupuncture point according the Traditional Chinese Medicine theory, besides, each patient was using 1-3 antihypertensive drug of a heterogeneous pharmacological group ranging from angiotensin-converting enzyme inhibitor (ACE inhibitor), diuretics, and beta blockers.

ELIGIBILITY:
Inclusion Criteria:

1. patient with isolated blood pressure diagnosis by physicians and BP >140/<90 mmHg
2. patient took the drug to control blood pressure for more than one year
3. age>65 years old
4. Willing to participate in this study

Exclusion Criteria:

1. Suspected acute stroke
2. chest pain or dyspnea
3. ingestion of short-acting antihypertensive medication within 2 h prior to the beginning of the study
4. body temperature >37.5∘C(99.5∘F)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-09-01 (Estimated); Study Completion 2019-05-31 (Estimated)

PRIMARY OUTCOMES:
blood pressure | change from Baseline Systolic Blood Pressure at 3 months
  measure blood pressure after the treatment compare the initial blood pressure

SECONDARY OUTCOMES:
Traditional Chinese Medicine constitution | use the questionnaire at Baseline, 1.5 month, and three month later
  use The Constitution in Chinese Medicine Questionnaire
heart rate variability | use ANS watch to monitor patient's condition at Baseline, 1.5 month, and three month later
  use autonomic nervous system (ANS) watch to monitor patient's heart rate variability, Low Frequency/High Frequency ratio

CONTACTS AND LOCATIONS:
Overall Officials: Kuei-Yu Huang, Study Director — Taipei City Hospital
Locations (1):
- Taipei City Hospital, Taipei, Taiwan